CLINICAL TRIAL: NCT07142239
Title: Comparative Analysis of Hematological Markers MPV, PLR, and NLR in Primary Versus Secondary Antiphospholipid Syndrome
Brief Title: Hematological Markers MPV, PLR, and NLR in Primary Versus Secondary Antiphospholipid Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Lecturer, New Valley University
Other Study IDs: HEM-APS
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Blood Cell Count; Mean Platelet Volume; Lymphocyte Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Primary APS
  Interventions: Diagnostic Test: • Complete blood count , MPV; Diagnostic Test: Calculation of PLR: Platelet count / Lymphocyte count and Calculation of NLR:; Diagnostic Test: Antiphospholipid antibody profile
- 2: secondary APS
  Interventions: Diagnostic Test: • Complete blood count , MPV; Diagnostic Test: Calculation of PLR: Platelet count / Lymphocyte count and Calculation of NLR:; Diagnostic Test: Antiphospholipid antibody profile

INTERVENTIONS:
Diagnostic Test: • Complete blood count , MPV — CBC report
Diagnostic Test: Calculation of PLR: Platelet count / Lymphocyte count and Calculation of NLR: — CBC report
Diagnostic Test: Antiphospholipid antibody profile — Patient record

SUMMARY:
Antiphospholipid syndrome is a thrombo-inflammatory autoimmune disorder with a complex antiphospholipid antibody-mediated pathogenesis, and high heterogeneity in clinical presentation and disease course. Clinical presentation in antiphospholipid syndrome includes venous and arterial thrombosis, pregnancy complications, and a broad range of microvascular and non-thrombotic manifestations

DETAILED DESCRIPTION:
APS may manifest as a primary, isolated condition or as a secondary disorder in conjunction with other autoimmune diseases, notably systemic lupus erythematosus (SLE) . The syndrome presents in two primary forms: thrombotic APS, marked by blood clots in both venous and arterial vessels, and obstetric APS (OAPS). While the criteria for APS diagnosis emphasize specific clinical and laboratory findings, recent research highlights the variability in antibody profiles and the potential for seronegative APS cases, complicating both diagnosis and management. Of note, thrombocytopenia is likely associated with more severe disease, and prolonged mild to moderate thrombocytopenia is linked to decreased long-term survival.

The neutrophil-lymphocyte ratio (NLR), defined as the ratio of the absolute value of neutrophils and lymphocytes in a peripheral venous blood stream, has been previously described as a non-invasive marker of the balance between the innate and adaptive immune response: neutrophils and lymphocytes are indeed indicators, respectively, of an active inflammatory state and of the regulatory pathway's activity in the immune system. Prior studies demonstrated that NLR is an easily available, cheap and widespread biomarker of systemic inflammation as well as a valid prognostic marker in multiple conditions, including cardiovascular, infectious, and chronic inflammatory diseases.

Alongside NLR, the platelet-to-lymphocyte ratio (PLR) has recently gained attention as a simple, cost-effective, and dependable marker that reflects inflammation, atherosclerosis, and cellular immune activation. An increased NLR, which represents the interaction between innate immunity driven mainly by neutrophils and adaptive immunity mediated by lymphocytes, and elevated PLR, as an indicator of inflammation and immune response, have been linked to acute thrombotic complications and are predictive of mortality in patients with solid tumors. However, their comparative evaluation between primary and secondary antiphospholipid syndrome (APS) remains limited.

Given the significant roles of inflammation, neutrophils, and platelets in the pathogenesis of venous thromboembolism (VTE), there has been growing interest in these parameters. NLR and PLR, both derived easily from complete blood counts, reflect primary hemostasis and inflammatory status. These ratios are minimally influenced by factors such as age, sex, and various physiological or pathological conditions, thereby potentially offering greater accuracy in detecting deep vein thrombosis (DVT) compared to other blood-based indices.

It is also noted that larger platelets are metabolically more active compared to smaller ones, producing higher quantities of β-thromboglobulin and thromboxane A2, substances associated with enhanced platelet activity, including increased expression of adhesion molecules and heightened aggregation ability.

NLR serves as an effective measure of systemic inflammation by reflecting the relative levels of neutrophils and lymphocytes. Substantial evidence now supports elevated NLR as a potential diagnostic and prognostic marker in a variety of cardiovascular and cerebrovascular diseases.

Similarly, PLR has been demonstrated to reliably reflect systemic inflammatory responses and is useful in predicting prognosis and outcomes in various conditions.

Mean platelet volume (MPV), which measures the average size of platelets in the blood, serves as an important parameter reflecting platelet function and activation, playing a key role in both inflammation and atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years)
* Diagnosis of APS based on updated Sydney classification criteria confirmed by: Clinical history of thrombosis and/or pregnancy morbidity, Persistent presence (≥12 weeks) of antiphospholipid antibodies (aCL, anti-β2-glycoprotein I, and/or lupus anticoagulant)

Exclusion criteria:

* Current infection or inflammatory condition unrelated to APS
* Hematological malignancies or other blood disorders
* Recent blood transfusion or platelet-altering medications other than APS treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be categorized as:
  Primary APS: APS without other systemic autoimmune diseases Secondary APS: APS associated with autoimmune diseases such as systemic lupus erythematosus (SLE)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-27 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
compare the levels and clinical implications of hematological markers mean platelet volume (MPV), platelet-to-lymphocyte ratio (PLR), and neutrophil-to-lymphocyte ratio (NLR) between patients diagnosed with primary APS and those with secondary APS | once
  comparison

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervera R, Serrano R, Pons-Estel GJ, Ceberio-Hualde L, Shoenfeld Y, de Ramon E, Buonaiuto V, Jacobsen S, Zeher MM, Tarr T, Tincani A, Taglietti M, Theodossiades G, Nomikou E, Galeazzi M, Bellisai F, Meroni PL, Derksen RH, de Groot PG, Baleva M, Mosca M, Bombardieri S, Houssiau F, Gris JC, Quere I, Hachulla E, Vasconcelos C, Fernandez-Nebro A, Haro M, Amoura Z, Miyara M, Tektonidou M, Espinosa G, Bertolaccini ML, Khamashta MA; Euro-Phospholipid Project Group (European Forum on Antiphospholipid Antibodies). Morbidity and mortality in the antiphospholipid syndrome during a 10-year period: a multicentre prospective study of 1000 patients. Ann Rheum Dis. 2015 Jun;74(6):1011-8. doi: 10.1136/annrheumdis-2013-204838. Epub 2014 Jan 24. PMID 24464962
- [Background] Shi Y, Zhao J, Jiang H, Huang C, Qi W, Song Y, Wang Q, Li M, Tian X, Zhao Y, Zeng X. Thrombocytopenia in primary antiphospholipid syndrome: association with prognosis and clinical implications. Rheumatology (Oxford). 2022 Dec 23;62(1):256-263. doi: 10.1093/rheumatology/keac264. PMID 35536236
- [Background] Garcia-Escobar A, Vera-Vera S, Tebar-Marquez D, Rivero-Santana B, Jurado-Roman A, Jimenez-Valero S, Galeote G, Cabrera JA, Moreno R. Neutrophil-to-lymphocyte ratio an inflammatory biomarker, and prognostic marker in heart failure, cardiovascular disease and chronic inflammatory diseases: New insights for a potential predictor of anti-cytokine therapy responsiveness. Microvasc Res. 2023 Nov;150:104598. doi: 10.1016/j.mvr.2023.104598. Epub 2023 Aug 24. PMID 37633337
- [Background] Farah R, Nseir W, Kagansky D, Khamisy-Farah R. The role of neutrophil-lymphocyte ratio, and mean platelet volume in detecting patients with acute venous thromboembolism. J Clin Lab Anal. 2020 Jan;34(1):e23010. doi: 10.1002/jcla.23010. Epub 2019 Sep 11. PMID 31508844
- [Background] Lattanzi S, Norata D, Broggi S, Meletti S, Switonska M, Slomka A, Silvestrini M. Neutrophil-to-Lymphocyte Ratio Predicts Early Neurological Deterioration after Endovascular Treatment in Patients with Ischemic Stroke. Life (Basel). 2022 Sep 10;12(9):1415. doi: 10.3390/life12091415. PMID 36143451
- [Background] Morkavuk SB, Kocaoz S, Korukluoglu B. Diagnostic value of Platelet/lymphocyte Ratio (PLR) for predicting sentinel axillary lymph node positivity in early-stage breast cancer compared with ultrasonography. Int J Clin Pract. 2021 Dec;75(12):e14939. doi: 10.1111/ijcp.14939. Epub 2021 Oct 12. PMID 34605138